CLINICAL TRIAL: NCT05610345
Title: The Effect of Placental Cord Drainage on Postpartum Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-08299-XP
Record Dates: First submitted 2022-10-26; First posted 2022-11-09 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Placenta Blood Drained Placenta Blood Not Drained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placenta Blood Drained (Experimental): Immediately after delayed cord clamping and cutting of the umbilical cord, the cord will be unclamped and blood with be drained until cessation of flow.
  Interventions: Procedure: Placental Blood Drainage
- Placenta Blood Not Drained (Active Comparator): This is the control group. The cord will not be unclamped.
  Interventions: Procedure: Placenta Blood Not Drained

INTERVENTIONS:
Procedure: Placental Blood Drainage — Immediately after vaginal delivery following delayed cord clamping and cutting of the cord, the cord will be unclamped and blood will be drained from the placenta until cessation of flow.
  Arms: Placenta Blood Drained
Procedure: Placenta Blood Not Drained — Placenta Blood Not Drained
  Arms: Placenta Blood Not Drained

SUMMARY:
To determine if placental cord drainage decreases the blood loss after spontaneous vaginal delivery

DETAILED DESCRIPTION:
Postpartum hemorrhage complicates 3% of pregnancies in the United States and is a leading cause of maternal morbidity and mortality. ACOG defines PPH as cumulative blood loss greater than 1000cc; however a blood loss >500cc should be considered abnormal. Primary PPH occurs in the first 24 hours and is largely secondary to uterine agony. ACOG as well as the WHO recommend active management of the third stage of labor to prevent PPH. This includes oxytocin administration, uterine massage, and gentle cord traction. Placental cord drainage (PCD) is the unclamping of the umbilical cord to allow for drainage of the blood from the placenta. It is another technique used to shorten the third stage of labor; however, it has not been well studied

ELIGIBILITY:
Inclusion Criteria:

* Singleton Gestation
* Ages 18-45
* English Speaking
* Third Trimester Gestation

Exclusion Criteria:

* Operative Vaginal Delivery
* Multiple Gestation
* Cesarean Delivery
* Episiotomy
* 3rd or 4th degree laceration
* Less than the Third Trimester of Pregnancy
* Chorioamnionitis
* History of Postpartum Hemorrhage
* Macrosomic Infant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Qualitative Blood Loss | Through delivery completion, on average 30 minutes
  Total Volume in Underbuttocks Drape - Initial Volume in Drape (amniotic fluid etc) + blood in laparotomy sponges

SECONDARY OUTCOMES:
Duration of Third Stage of Labor | On average 30 minutes
  After neonatal delivery to delivery of the placenta
Retained Placenta | 30 minutes after delivery
  Placenta not delivered > 30 minutes
Postpartum Hemorrhage | 30 minutes to 1 hour after delivery
  Blood Loss Greater than 1000cc
Blood Loss > 500 cc | 30 minutes to 1 hour after delivery
  Greater than average postpartum blood loss
Need for Blood Transfusion | Up to 24 hours postpartum
  In event of HgB <7 or active bleeding
Percent Drop in HgB and Hct | Up to 48 hours following delivery
  Lab draw following delivery
Additional Uterotonic Administration | 30 minutes to 1 hour following delivery
  Medications administered to stop postpartum bleeding
Endometritis | Up to 12 weeks following delivery
  Infection of myometrium of uterus

CONTACTS AND LOCATIONS:
Overall Officials: John Schorge, MD, FACS, Study Chair — Regional One Health
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] WHO recommendations on maternal health: guidelines approved by the WHO Guidelines Review Committee [Internet]. Geneva: World Health Organization; 2017. Available from http://www.ncbi.nlm.nih.gov/books/NBK615100/ PMID 40455892
- [Result] Roy P, Sujatha MS, Bhandiwad A, Biswas B, Chatterjee A. Placental Blood Drainage as a Part of Active Management of Third Stage of Labour After Spontaneous Vaginal Delivery. J Obstet Gynaecol India. 2016 Oct;66(Suppl 1):242-5. doi: 10.1007/s13224-016-0857-3. Epub 2016 Mar 12. PMID 27651611
- [Result] Wu HL, Chen XW, Wang P, Wang QM. Effects of placental cord drainage in the third stage of labour: A meta-analysis. Sci Rep. 2017 Aug 1;7(1):7067. doi: 10.1038/s41598-017-07722-7. PMID 28765609
- [Result] Vasconcelos FB, Katz L, Coutinho I, Lins VL, de Amorim MM. Placental cord drainage in the third stage of labor: Randomized clinical trial. PLoS One. 2018 May 2;13(5):e0195650. doi: 10.1371/journal.pone.0195650. eCollection 2018. PMID 29718920